CLINICAL TRIAL: NCT02940912
Title: Double Bind Randomized Placebo-controlled Cross-over Study to Evaluate Effect of Continuous Apomorphine During the Night on Sleep Disorders in Insomniac Patients With Parkinson's Disease
Brief Title: Effect of Continuous Apomorphine During the Night on Sleep Disorders in Insomniac Patients With Parkinson's Disease
Acronym: APOMORPHEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-005793-37
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Insomnia; Sleep disorders; Polysomnography; Apomorphine; Multiple sleep latency test; Parkinson Disease Sleep Scale 2 (PDSS-2)
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apomorphine (5 mg/ml) (Active Comparator): Active phase is apomorphine (from 0.5 mg (0.1 ml) to maximum 5 mg (1 ml)/hour of apomorphine), delivered with a pump (subcutaneous administration), during 22 days.
  Interventions: Drug: Apomorphine
- Physiologic serum (Placebo Comparator): Physiological serum (from 0.1 ml to maximum 1 ml/ hour), delivered with a pump (subcutaneous administration), during 22 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine — cross-over with start with Apokinon in the 1st phase- in the 2nd phase of continuous treatment with Physiologic Serum.
  Other Names: Apokinon
  Arms: Apomorphine (5 mg/ml)
Drug: Placebo — cross-over with start with.Physiologic Serum in the 1st phase- in the 2nd phase of continuous treatment with Apokinon.
  Other Names: Physiologic Serum
  Arms: Physiologic serum

SUMMARY:
The purpose of the study is to demonstrate that continuous apomorphine treatment during the night compared with placebo improves sleep quality in insomniac patient with Parkinson's disease.

DETAILED DESCRIPTION:
Sleep disorders are very common in Parkinson's disease (PD). They are present in almost all patients. They have an important impact on quality of life. To improve the comfort of patients, neurologists typically offer either dispersible form of levodopa, prolonged release dopaminergic agonists treatments or deep brain stimulation surgery. Unfortunately these treatments are too short-acting for the dispersible form of levodopa or not always sufficient for the oral or transdermal dopamine agonist or are very heavy to implement as surgery.

Some sleep disorders such as restless legs syndrome and periodic leg movements, and obstructive sleep apnoea syndrome, seem to be more frequent in PD patients than in general population and could be improved by a continuous dopaminergic treatment the night.

Finally, daytime sleepiness is a major problem in PD patients. Although it seems most often linked to dopaminergic treatments given during the day, it could also be, in some patients the result of a very bad night's sleep, leading to a rebound of sleep during the day.

The main objective is to demonstrate that compared with placebo, nocturnal continuous apomorphine treatment improves sleep quality assessed by the patient on the PDSS-2 scale in fluctuating parkinsonian patients with complaints of insomnia.

The secondary objectives are to measure the effectiveness of nocturnal continuous apomorphine on sleep quality : total sleep time, sleep efficiency, arousal index, ventilatory events and legs movements indexes, to measure the relative proportion of sleep stages (N1, N2, N3, Rapid Eye Movement ou REM sleep), position changes during sleep index and the percentage of time spent in the supine position, percentage of time with SpO2 <90%), sleepiness (Epworth and Multiple Sleep Latency Test) and their consequences on quality of life (EuroQol 5), depressive symptoms (Beck II), anxiety (STAI), overall cognition (MOCA), pain and engine condition after waking up.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease ( Hughes AJ et al. 2001)
* Patients with motor fluctuations
* Chronic Insomnia disorder criteria according to the criteria of DMS- V ( American Psychiatric Association, 2013) and insomnia severity index > 15
* Able to use independently the device required for treatment by apomorphine
* Collection of written informed consent (legal obligation for any project under the public health law , bioethics laws and / or CNIL) .
* Affiliate to social security or beneficiary of such a regime

Exclusion Criteria:

* Atypical Parkinsonian Syndromes
* Parkinson's disease with dementia (Montreal Cognitive Assessment (MoCA) <25/30 (NASREDDINE and al., 2012))

  * Parkinson's disease with hallucinations
  * Parkinson's disease with impulse Control disorder (ICD)
  * Parkinson's disease already treated with APOMORPHINE pump or justifying the use of the pump continuously day and night
  * Another obvious severe disease explaining insomnia
  * Exclusion for monitoring difficulties (mutation, insufficient motivation, priority associated pathology in care)
  * Patient unwilling to accept a pump
  * Patient not accepting polysomnography and multiple sleep latency test
  * Patient with health problems or a skin disease precluding continuous subcutaneous infusion
  * Female parturient or nursing
  * Cardiac dysrhythmia precluding treatment with domperidone or apomorphine (increased QTc ≥ 440 ms in men, QTc ≥ 450 ms in women)
  * Treatments forbidden in association with apomorphine such as:

    * antiemetic neuroleptics
    * Tetrabenazine
  * Excessive alcohol consumption
  * Contraindications for apomorphine:

    * Hypersensitivity to apomorphine or one of the excipients
    * Respiratory Depression
    * Hepatic impairment
    * Intellectual Disability
    * Dementia

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline PDSS2 score (Parkinson's Disease Sleep Scale) at the end of the sequence | 53 days
  This score is a score range, it's the difference between PDSS2 score at day18 and day 1 (for the first sequence) and difference between day 53 and day 36 (for the second sequence).

SECONDARY OUTCOMES:
Total sleep time period | 53 days
  Variable will be measured from the polysomnography recordings
Total sleep time (non-Rapid Eye Movements (REM) stages 1,2,3 plus REM sleep) | 53 days
  Variables will be measured from the polysomnography recordings
Length of the intra-sleep wakefulness | 53 days
Sleep efficiency (total sleep time based on the total sleep period) | 53 days
Duration of each sleep stage of the total sleep time | 53 days
Subjective sleepiness on the Epworth Sleepiness Scale | 53 days
Sleep latency (between light extinction and the first period of sleep) | 53 days
Arousal index | 53 days
Apnea / hypopnea Index | 53 days
Percentage of time spent with a saturation below 90% | 53 days
Periodic leg movement index | 53 days
Percentage of REM sleep time with tonic and phasic activity | 53 days
Objective sleepiness on Multiple Sleep Latency Test | 53 days

CONTACTS AND LOCATIONS:
Overall Officials: Valérie COCHEN DE COCK, PI, MD, PhD, Principal Investigator — Clinique BEAU SOLEIL, 34070 Montpellier; Emmanuel FLAMAND-ROZE, PI, MD, PhD, Principal Investigator — Hopital PITIE-SALPETRIERE, 75013 Paris
Locations (9):
- France (9):
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Hôpital de la TIMONE, Marseille
  - Clinique Beau Soleil, Montpellier
  - CHU de NANTES - HOPITAL NORD, Nantes
  - CHU de NIMES, Nîmes
  - Chu Ponchaillou, Rennes
  - Hôpital CIVIL, Strasbourg
  - Hôpital de HAUTEPIERRE, Strasbourg
  - Centre hospitalier JACQUES LACARIN, Vichy

REFERENCES:
- [Derived] De Cock VC, Dodet P, Leu-Semenescu S, Aerts C, Castelnovo G, Abril B, Drapier S, Olivet H, Corbille AG, Leclair-Visonneau L, Sallansonnet-Froment M, Lebouteux M, Anheim M, Ruppert E, Vitello N, Eusebio A, Lambert I, Marques A, Fantini ML, Devos D, Monaca C, Benard-Serre N, Lacombe S, Vidailhet M, Arnulf I, Doulazmi M, Roze E. Safety and efficacy of subcutaneous night-time only apomorphine infusion to treat insomnia in patients with Parkinson's disease (APOMORPHEE): a multicentre, randomised, controlled, double-blind crossover study. Lancet Neurol. 2022 May;21(5):428-437. doi: 10.1016/S1474-4422(22)00085-0. PMID 35429481